CLINICAL TRIAL: NCT03287648
Title: Simultaneous Spectral-domain Optical Coherence Tomography and Blue-fundus Autofluorescence in Eyes With Alteration of the Foveal Contour
Brief Title: Simultaneous OCT and B-FAF in Eyes With Alteration of the Foveal Contour
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Molise (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Roberto dell'Omo, Associate Professor, University of Molise
Other Study IDs: 0004/2017
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Lamellar Macular Hole; Lamellar Macular Pseudohole
Keywords: optical coherence tomography; blue fundus autofluorescence
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: optical coherence tomography and blue-fundus autofluorescence — Simultaneous infra-red and optical coherence tomography (cube and radial pattern) centered on the fovea Simultaneous fundus autofluorescence and optical coherence tomography (radial pattern) centered on the fovea
  Other Names: infra-red, color pictures

SUMMARY:
Some alterations of the foveal contour do not meet the criteria established for the definition of lamellar macular hole on the basis of optical coherence tomography (OCT). However, these alterations may show an appearance, on blue fundus autofluorescence (B-FAF) imaging, reminiscent of lamellar macular hole.

The aim of the study is to evaluate in detail these alterations recording simultaneously OCT and B-FAF.

DETAILED DESCRIPTION:
All images will be collected using the Heidelberg Spectralis system (Heidelberg Engineering, Heidelberg, Germany) according to the prespecified imaging protocols. Blue-fundus autofluorescence (excitation wavelength at 488 nm and barrier filter at 500 nm) images and SD-OCT images will be obtained after pupil dilation.

The OCT recording protocol will consist of a sequence of 37 horizontal sections, spaced 120-µm apart, covering an area of 20° or 30° horizontally by 15° vertically, and a sequence of 24 radial sections recorded in the high-resolution (HR) mode simultaneously with infrared (IR) images.

In addition, simultaneous B-FAF/OCT images will be acquired (horizontal, and vertical OCT sections, centered on the fovea and recorded in the HR mode).

The same OCT/FAF protocol will be used for the study eye and for the fellow eye.

For the study eyes that had been examined in the past, the ''Follow-up'' function will be used in addition to the prespecified protocol to evaluate if any changes had occurred since the last scan.

Multiple other morphological characteristics will be analyzed using OCT imaging, including the status of the posterior cortex, the presence of operculum, the integrity/disruption of the external limiting membrane (ELM), ellipsoid zone (EZ), and the central and minimal foveal thickness (CFT and mFT respectively). The latter will be defined as the thinnest part of the fovea within the foveal pit identified by examining radial scans whereas the former will be measured in relation to the highest point of the foveal bulge.

All measurements will be performed using the Spectralis built-in manual caliper function at high magnification after adjusting the scale to 1:1 µm except for CFT, which will be calculated using the automated ''thickness map'' function of the Heidelberg Eye Explorer.

ELIGIBILITY:
Inclusion Criteria:

* alteration of the foveal contour not classifiable as lamellar or pseudo macular hole
* focal, well-defined increased autofluorescence signal at the fovea

Exclusion Criteria:

* intraretinal cysts not associated with break of the inner retina
* juxtafoveal telangiectasia
* ring of increased B-FAF
* vitelliform and pseudovitelliform lesions
* history of diabetes, retinal vein occlusion, uveitis, CSR, AMD or any other retinal -disease potentially associated with intra or subretinal fluid
* macular drusen
* history of submacular hemorrhage

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients affected by alteration of the foveal contour associated with increased autofluorescence signal at the fovea
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Relationship between OCT and B-FAF findings | 6 months
  Measurements of the diameters of the holes expressed in microns, on OCT and B-FAF images respectively, will be collected. The topographic correlation between the area of increased B-FAF signal and the corresponding area on OCT, will be examined.

SECONDARY OUTCOMES:
Relationship between OCT and B-FAF characteristics and logMAR visual acuity | 6 months
  The relationship between central foveal thickness and logMAR visual acuity will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- University of Molise, Campobasso, Italy

IPD SHARING:
Plan to Share IPD: Undecided